CLINICAL TRIAL: NCT02193464
Title: Observational Study Using Inflammatory Bowel Disease Registry in Daegu-Gyeongbuk, Southeastern Area of Korea
Brief Title: Inflammatory Bowel Disease Registry in Daegu-Gyeongbuk
Acronym: EPICODE
Status: Recruiting | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Collaborators: Yeungnam University Hospital (Other); Daegu Catholic University Medical Center (Other); DongGuk University (Other)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Professor, Kyungpook National University Hospital
Other Study IDs: EPICODE
Record Dates: First submitted 2014-07-16; First posted 2014-07-17 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Idiopathic Chronic Inflammatory Bowel Disease
Keywords: inflammatory bowel disease, registry, incidence, Korea
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- inflammatory bowel disease

SUMMARY:
The purpose of this study is to investigate the incidence and natural course of inflammatory bowel disease in the southeastern area of Korea.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of inflammatory bowel disease including Crohn's disease and ulcerative colitis
* Followed up for at least 6 months for the correct diagnosis

Exclusion Criteria:

* Patients who do not live in Daegu-Gyeongbuk province

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with inflammatory bowel disease from primary, secondary, and tertiary hospital in Daegu-Gyeongbuk province of Korea.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
All newly diagnosed cases | one year
  In one year, all inflammatory bowel disease including Crohn's disease and ulcerative colitis which is newly diagnosed in Daegu-Gyeongbuk province of Korea is recorded.

SECONDARY OUTCOMES:
All operation cases | one year
  For one year, all patients who have surgical managements for IBD are counted.

OTHER OUTCOMES:
All cases of disease relapse | one year
  For one year, all patients who have disease worsening are counted.

CONTACTS AND LOCATIONS:
Overall Officials: Eun Soo Kim, MD, PhD, Principal Investigator — Keimyung University School of Medicine
Locations (1):
- Keimyung University Dongsan Medical Center, Daegu, South Korea